Version: 2.0 Version Date: 2024/2/1

## Ultrasound-assisted vs. real-time ultrasound-guided paracentral approach combined lumbar and epidural anesthesia in elderly patients: a randomized controlled study

Version: 2.0

Version Date: 2024/2/1

## Statistical analysis

All statistical analysis were performed using Statistical Package for Social Sciences (SPSS) for Windows software version 23. Numerical variables were expressed as mean  $\pm$  SD or median (minimum–maximum). Categorical variables were expressed as frequency (%). Test of normality was done using Kolmogorov–Smirnov test. One-Way analysis of variance (ANOVA) was used to compare means if data distribution was normal, or nonparametric test Mann-Whitney U was used if data was not distributed normally. Pearson chi-square or Fischer's exact test was used for assessing categorical variables. Log rank test was used to evaluate the time difference in the first administration of diclofenac sodium after surgery, and hazard ratio (HR) was used to evaluate the benefit. All tests were two-tailed, and the significance level was set at  $\alpha$  0.05.